CLINICAL TRIAL: NCT04882878
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Nipocalimab in Adult Participants With Active Systemic Lupus Erythematosus
Brief Title: A Study of Nipocalimab in Adult Participants With Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109011; 80202135SLE2001 (Other: Janssen Research & Development, LLC); 2020-005569-14 (EudraCT Number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; SLE; Nipocalimab; Lupus SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Placebo (Placebo Comparator): Participants will receive placebo intravenously (IV) every two weeks (q2w) through Week 50 along with standard-of-care treatments (that is, immunomodulators, antimalarial drugs and Glucocorticoids [GCs]).
  Interventions: Other: Placebo; Drug: Standard-of-care treatment
- Group 2: Nipocalimab Dose 1 (Experimental): Participants will receive nipocalimab dose 1 intravenously (IV) q2w through Week 50 along with standard-of-care treatments (that is, immunomodulators, antimalarial drugs and GCs).
  Interventions: Drug: Nipocalimab; Drug: Standard-of-care treatment
- Group 3: Nipocalimab Dose 2 (Experimental): Participants will receive nipocalimab dose 2 intravenously (IV) q2w through Week 50 along with standard-of-care treatments (that is, immunomodulators, antimalarial drugs and GCs).
  Interventions: Drug: Nipocalimab; Drug: Standard-of-care treatment

INTERVENTIONS:
Other: Placebo — Placebo will be administered intravenously.
  Arms: Group 1: Placebo
Drug: Nipocalimab — Nipocalimab dose 1 and dose 2 will be administered intravenously.
  Other Names: JNJ-80202135; M281
  Arms: Group 2: Nipocalimab Dose 1; Group 3: Nipocalimab Dose 2
Drug: Standard-of-care treatment — Standard-of-care treatment including immunomodulators, antimalarial drugs and GCs will be administered orally.

SUMMARY:
The purpose of this study is to evaluate the efficacy of nipocalimab versus placebo in participants with active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
SLE is a complex, immune-mediated inflammatory disorder of unknown etiology that can affect almost any organ system and follows a waxing and waning disease course. In SLE, the immune system attacks the body cells and tissues and the resulting inflammation and tissue damage can harm the heart, joints, skin, lungs, blood vessels, liver, kidneys, and nervous system. Nipocalimab is a fully human aglycosylated immunoglobulin (Ig)G1 monoclonal antibody designed to selectively bind, saturate, and block the IgG binding site on the endogenous neonatal fragment crystallizable receptor (FcRn). Thus, nipocalimab, a FcRn antibody, has potential in treatment of SLE through lowering of pathogenic IgGs and immune complexes. The study will consist of a Screening Period (less than or equal to [<=] 6 Weeks), double-blind Treatment Period (52 Weeks), and a Follow-up Period (6 Weeks). Key safety assessments will include adverse events (AEs), serious adverse events (SAEs), adverse events of special interests (AESIs), clinical laboratory tests (hematology, chemistry, urinalysis, and lipid profile) and vital signs. The total duration of the study is up to 64 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of systemic lupus erythematosus (SLE) greater than or equal to (>=) 6 months prior to the screening visit and according to Systemic Lupus International Collaborating Clinics (SLICC)-2012 classification criteria: at least 4 criteria fulfilled, with at least 1 clinical criterion and 1 immunologic criterion
* Has at least 1 BILAG (british isles lupus assessment group) A and/or 2 BILAG B scores observed during screening
* Must have at least moderately active SLE, as defined as systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score >= 6 at screening visit. Must also have SLEDAI 2K >= 4 for clinical features (that is, SLEDAI-2K score excluding headache and laboratory abnormalities) present at Week 0 prior to randomization
* Has a CLASI (cutaneous lupus erythematosus disease area and severity index) activity score of at least 6 (excluding diffuse non-inflammatory alopecia) or at least 4 joints with pain and signs of inflammation (active joints) at screening or at Week 0, or both
* At least 1 unequivocally positive autoantibody test including antinuclear antibodies (ANA) (>= 1:80) and/or anti-double stranded deoxyribonucleic acid (dsDNA) antibodies (level >= 75 international units/milliliter [IU/mL]) and/or anti-Smith antibodies (>120 Absorbance unit/milliliter [AU/mL]) detected during screening
* Must be receiving 1 or more of the following protocol-permitted, systemic standard-of-care treatments prior to first administration of study intervention at a stable dose: oral glucocorticoids, antimalarial or up to 2 immunomodulatory drugs

Exclusion Criteria:

* Current or history of, severe, progressive, or uncontrolled renal disease, with the exception of active lupus nephritis (LN). Have severe active LN as determined by sponsor (or designee) adjudication. Control of renal disease must be documented with at least 2 measurements of proteinuria or urine protein/creatinine ratio (UPCR) over the 6 months prior to screening
* Has any unstable or progressive manifestation of SLE that is likely to warrant escalation in therapy beyond permitted background medications
* Confirmed or suspected inflammatory diseases that might confound the evaluations of efficacy
* Has a severe infection including opportunistic infections requiring parenteral anti-infectives, and/or hospitalization within 8 weeks prior to screening
* Has received a single B-cell targeting agent within 3 months prior to first administration of study intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving an Systemic Lupus Erythematosus (SLE) Responder Index (SRI)-4 Composite Response at Week 24 | Week 24
  SLE SRI-4 composite response is a composite of at least 4-point improvement in SLE Disease Activity Index 2000(SLEDAI-2K), no worsening in British Isles Lupus Assessment Group (BILAG), no worsening in Physician's Global Assessment of Disease Activity score (PGA) and not meeting study treatment failure criteria.

SECONDARY OUTCOMES:
Percentage of Participants with Baseline Active Mucocutaneous Lupus Manifestations (Cutaneous Lupus Erythematosus Disease Area and Severity Index [CLASI] Activity Score >= 6) Achieving >= 50 Percent (%) Reduction in the CLASI Activity Score at Week 24 | Week 24
  Percentage of participants achieving at least 50% improvement in CLASI Activity Score at Week 24 will be reported in participants with a CLASI Activity Score of 6 or greater at baseline. Cutaneous lupus disease activity and severity will be measured by the CLASI. The CLASI is an instrument to assess the disease activity and damage caused to the skin for cutaneous lupus erythematosus participants with or without systemic involvement. The CLASI consists of 2 scores; the first summarizes the activity of the disease while the second is a measure of the damage caused by the disease.
Percentage of Participants with Baseline Arthritis (with at Least 4 Active Joints at Baseline) Achieving >= 50% Reduction in Active Joints at Week 24 | Week 24
  Percentage of participants with baseline arthritis (with at least 4 active joints at baseline) achieving >= 50% reduction in active joints at Week 24 will be reported.
Percentage of Participants with >= 4 Point Improvement in SLE Disease Activity Index 2000 (SLEDAI-2K) at Week 24 | Week 24
  Percentage of participants achieving at least 4 point improvement in SLEDAI-2K will be reported. The SLEDAI-2K is an established, validated SLE activity index. It is based on the presence of 24 features in 9 organ systems and measures disease activity in SLE participants at the time of the visit or in the previous 30 days; the index is weighted according to the feature. Features are scored by the assessing physician if present at the time of the visit or within the last 30 days, with more severe features having higher scores, and then simply added to determine the total SLEDAI-2K score, which ranges from 0 to 105, with higher scores representing increased disease activity.
Percentage of Participants Achieving the British Isles Lupus Assessment Group (BILAG) Composite Lupus Assessment (BICLA) Response at Week 24 | Week 24
  Percentage of participants achieving BICLA Response (BILAG-2004 disease activity improvement without worsening, and without worsening of SLEDAI-2K or PGA compared to baseline) at Week 24 will be reported.
Time to First Flare Through Week 24 | Up to Week 24
  Time to first flare through Week 24, with flare defined as either 1 or more new BILAG A or 2 or more new BILAG B scores will be reported.
Percentage of Participants Achieving SRI-4 Composite Response at Week 52 | Week 52
  Percentage of participants achieving SRI-4 composite response at Week 52 will be reported.
Percentage of Participants Receiving >= 10 milligram/day (mg/day) Prednisone or Equivalent at Baseline who Achieve Week 6-16 Glucocorticoid (GC) Taper Goal (at Week 16 to <= 7.5 mg/day Prednisone or Equivalent) and Maintain that Reduction Until Week 24 | Up to Week 24
  Percentage of participants receiving >= 10 mg/day prednisone or equivalent at baseline who achieve Week 6-16 GC taper goal (at Week 16 to <= 7.5 mg/day prednisone or equivalent) and maintain that reduction until Week 24 will be reported.
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) Through Week 58 | Up to Week 58
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Treatment-emergent Serious Adverse Events (SAEs) Through Week 58 | Up to Week 58
  SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. Treatment-emergent SAEs are defined as SAEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Treatment-emergent Adverse Events of Special interests (AESIs) Through Week 58 | Up to Week 58
  Percentage of participants with treatment-emergent AESIs will be reported. Treatment-emergent adverse events associated with the following situations are considered as AESIs: infections that are severe or require intravenous anti-infective or operative/invasive intervention, hypoalbuminemia with albumin less than (<) 20 gram/liter (g/L) (<2.0 gram/deciliter [g/dL]).
Percentage of Participants with Treatment-emergent AEs leading to treatment discontinuation Through Week 58 | Up to Week 58
  Percentage of participants with treatment-emergent AEs leading to discontinuation of study intervention will be reported.
Number of Participants with Change from Baseline in Laboratory Parameters Over Time | Up to Week 58
  Number of participants with change from baseline in laboratory parameters (hematology, chemistry, urinalysis and lipid profile) over time will be reported.
Number of Participants with Change from Baseline in Vital Signs Parameters Over Time | Up to Week 58
  Number of participants with change from baseline in vital sign parameters (temperature, pulse/heart rate, respiratory rate, and blood pressure) will be reported.
Serum Concentration of Nipocalimab Over Time | Up to Week 58
  Serum concentrations of nipocalimab over time in participants receiving active study intervention will be reported.
Number of Participants with Antibodies to Nipocalimab (Anti-Drug Antibodies [ADAs] and Neutralizing Antibodies [Nabs]) | Up to Week 58
  Number of participants with antibodies to nipocalimab (ADAs and Nabs) in participants receiving active study intervention will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (86):
- United States (21):
  - Valerius Medical Group & Research Center, Los Alamitos, California
  - Desert Medical Advances, Rancho Mirage, California
  - Wolverine Clinical Trials, Santa Ana, California
  - Millennium Clinical Trials LLC, Westlake Village, California
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - GNP Research, Cooper City, Florida
  - South Coast Research Center, Miami, Florida
  - Advanced Clinical Research of Orlando, Ocoee, Florida
  - Omega Research Consultants, Orlando, Florida
  - Millennium Research, Ormond Beach, Florida
  - North Georgia Rheumatology, PC, Lawrenceville, Georgia
  - Atlanta Research Center for Rheumatology, Marietta, Georgia
  - West County Rheumatology, St Louis, Missouri
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Paramount Medical Research & Consulting, Middleburg Heights, Ohio
  - Dr. Ramesh Gupta, Memphis, Tennessee
  - Arthritis and Rheumatology Research Institute, Allen, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - Epic Medical Research, Red Oak, Texas
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Argentina (8):
  - Centro Médico Reumatológico (OMI), Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - ARCIS Salud SRL Aprillus asistencia e investigacion, CABA
  - Clinica Adventista Belgrano, Ciudad de Buenos Aires
  - Hospital Italiano La Plata, La Plata
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto de Reumatologia - Ir Medical Center S.A., Mendoza
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Diagnostic-Consultative Center (DCC) Aleksandrovska, Sofia
  - UMHAT St. Ivan Rilski, Sofia
- Colombia (5):
  - Clinica de la Costa SAS, Barranquilla
  - Centro de Investigacion Medico Asistencial SAS - CIMEDICAL SAS, Barranquilla
  - Centro de Investigación en Reumatología y especialidades médicas S.A.S. - CIREEM S.A.S., Bogotá
  - Servimed S A S, Bucaramanga
  - IPS Preventive Care SAS, Chía
- Germany (2):
  - Praxis Dr. med. Beate Schwarz - Germany, Langenau
  - Universitaetsklinikum Leipzig, Leipzig
- Hungary (3):
  - Betegapolo Irgalmas Rend Budai Irgalmasrendi Korhaz, Budapest
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Belvarosi Egeszseghaz Kft. (Leda-Platan Maganklinika es Sebeszeti Kozpont), Zalaegerszeg
- Japan (12):
  - National Hospital Organization Chiba East Hospital, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - National Center for Global Health and Medicine Kohnodai hospital, Ichikawa
  - St Marianna University Hospital, Kanagawa
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Osaka Metropolitan University Hospital, Osaka
  - Tohoku University Hospital, Sendai
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - St. Luke's International Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - University of Tsukuba Hospital, Tsukuba
- Poland (10):
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz
  - Nzoz Bif Med, Bytom
  - Malopolskie Badania Kliniczne Sp z o o, Krakow
  - Centrum Medyczne Plejady, Krakow
  - NZOZ Lecznica MAK MED S C, Nadarzyn
  - Twoja Przychodnia Poznanskie Centrum Medyczne, Poznan
  - AI Centrum Medyczne, Poznan
  - Prywatna Praktyka Lekarska Prof Um Dr Hab Med Pawel Hrycaj, Poznan
  - Uniwersytecki Szpital Kliniczny w Rzeszowie, Rzeszów
  - MICS Centrum Medyczne Warszawa, Warsaw
- South Africa (3):
  - Panorama Medical Centre, Cape Town
  - Excellentis Clinical trial Consultants, George
  - Winelands Rheumatology Centre, Stellenbosch
- Spain (5):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. de Navarra, Pamplona
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taipei Medical University, Taipei
- Ukraine (10):
  - Municipal Non-Profit Enterprise 'Chernihiv Regional Hospital' of Chernihiv Regional Council, Chernihiv
  - Municipal Non-Profit Enterprise of Kharkiv Regional Council 'Regional Clinical Hospital', Kharkiv
  - Medical Center 'Ok Clinic' of International Institute of Clinical Research LLC, Kyiv
  - Medbud-Clinic LLC, Kyiv
  - Kyiv Railway Clinical Hospital #2 Of Branch 'Health Center' Of The Company 'Ukrainian Railway', Kyiv
  - Medical Center 'Consylium Medical', Kyiv
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - ME Poltava Regional Clinical Hospital named after M.V. Sklifosovsky of Poltava Regional Consuil, Poltava
  - MNPE 'Vinnytsia Regional Clinical Hospital named after M.I. Pyrogov of Vinnytsia Regional Council', Vinnytsia
  - Medical Center LLC 'Modern Clinic', Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency